CLINICAL TRIAL: NCT05561296
Title: Safety and Efficacy of Astigmatism Correction by Iris-registration Guided Corneal Relaxing Incisions or Toric IOL Implantation During Femtosecond Laser-assisted Cataract Surgery
Brief Title: Astigmatism Management With Iris-registration Guided Corneal Relaxing Incisions or Toric IOLs During Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kenneth J Rosenthal (Other)
Collaborators: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Kenneth J Rosenthal, Sponsor-Investigator, Rosenthal Eye Surgery
Organization: Rosenthal Eye Surgery (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KJR/2022/01
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Astigmatism; Cataract
Keywords: corneal relaxing incisions; toric IOL; iris registration; femtosecond laser-assisted cataract surgery
MeSH Terms: conditions — Astigmatism; Cataract

STUDY DESIGN:
Intervention Model Description: This prospective, open-label, single-center, non-randomized, interventional study will include 50 patients who will undergo femtosecond laser-assisted cataract surgery (Catalys) and astigmatism correction by either EyHance toric II IOLs or corneal relaxing incisions and implantation of EyHance IOL. The alignment would be guided by preoperatively obtained iris registration using Cassini Ambient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Astigmatism correction with iris registration guided corneal relaxing incisions (Other): This sub-group will include patients who will undergo femtosecond laser-assisted cataract surgery (Catalys) and astigmatism correction using corneal relaxing incisions and implantation of EyHance IOL. The alignment would be guided by preoperatively obtained iris registration using Cassini Ambient.
  Interventions: Procedure: Femtosecond laser assisted cataract surgery with astigmatism management
- Astigmatism correction with iris registration guided implantation of toric IOLs (Other): This sub-group will include patients who will undergo femtosecond laser-assisted cataract surgery (Catalys) and astigmatism correction with the implantation of EyHance toric II IOLs. The alignment would be guided by preoperatively obtained iris registration using Cassini Ambient.
  Interventions: Procedure: Femtosecond laser assisted cataract surgery with astigmatism management

INTERVENTIONS:
Procedure: Femtosecond laser assisted cataract surgery with astigmatism management — The alignment would be guided by preoperatively obtained iris registration using Cassini Ambient. Patients will undergo femtosecond laser-assisted cataract surgery with Catalys femtosecond laser.

SUMMARY:
Most of the patients presenting for cataract surgery also have pre-existing corneal astigmatism which if left uncorrected can adversely affect visual and refractive outcomes after cataract surgery. Pre-existing astigmatism at the time of cataract surgery can be corrected by either corneal relaxing incisions or implantation of toric IOLs. While the safety and efficacy of these procedures are well established, there are various challenges associated with these techniques that surgeons need to overcome to achieve good outcomes postoperatively.

The use of iris registration technology that automatically compensates for cyclotorsion has the potential to improve the alignment accuracy of CRI or toric IOLs. The Cassini Ambient and Catalys Femtosecond Laser incorporate this technology to help cataract surgeons accurately align toric IOLs on the intended axis of implantation or accurately place CRI on the intended meridian. The present study is aimed at evaluating the efficacy of astigmatism correction during femtosecond laser-assisted cataract surgery with Catalys femtosecond laser. The patients will either undergo iris registration guided CRIs or iris registration guided alignment of toric IOLs.

DETAILED DESCRIPTION:
Surgical correction of astigmatism using corneal relaxing incisions or toric IOLs have been widely adopted to correct pre-existing astigmatism in cataract surgery patients. While the safety and efficacy of these procedures are well established, there are various challenges associated with these techniques that surgeons need to overcome to achieve good outcomes postoperatively; for instance, correction of astigmatism either with corneal relaxing incisions (CRIs) or toric IOLs during cataract surgery requires appropriate pre-operative planning based on corneal curvature measurements, biometry, nomogram/IOL selection, accurate marking for the placement of CRI/implantation of toric IOL on the intended axis, intraoperative alignment, cyclotorsion compensation, and postoperative IOL rotation, etc.

The Cassini Ambient and Catalys Femtosecond Laser incorporate this technology to help cataract surgeons accurately align toric IOLs on the intended axis of implantation or accurately place CRI on the intended meridian. This is expected to improve patients' visual functioning and reduce spectacle dependence postoperatively. The Cassini Ambient provides the preoperative anterior and posterior astigmatism with iris registration. The new Catalys Precision Laser System (Johnson & Johnson Vision) with cOS 6.0 software facilitates direct importation of preoperative data from the Cassini via a wireless connection or USB drive, eliminates the need for manual axis marking as it compares the pre- and intra-operative iris anatomy data and compensates for tilt and rotation so that the laser marks are perfectly aligned to the steep meridian and the target axis. Linking preoperative diagnostic information to the laser minimizes data entry and transcription errors. It also eliminates several steps in the planning process for toric IOLs and CRI, thus improving the overall accuracy of the astigmatism correction procedure and reducing chances for error.

ELIGIBILITY:
Inclusion Criteria:

* Patients desirous of undergoing cataract surgery.
* Pre-existing corneal astigmatism requiring either CRIs or toric IOL implantation.
* Patients in whom iris registration link between Cassini Ambient and Catalys femtosecond laser is successful.

Exclusion Criteria:

Patients will be excluded from participating in the study due to any of the following reasons:

* Insufficient pupil dilation to complete Catalys treatment
* Clinically significant corneal pathology precluding reliable Cassini topographical measurement of any cause
* Preoperative corneal astigmatism greater than 4.00 D, or astigmatism requiring both CRIs and implantation of toric intraocular lens for correction.
* Cassini topographical measurement deemed inconsistent with historical topographies and refractive error based on clinical judgment
* Visually significant ocular surface disease (OSD) precluding reliable measurements and/or anticipated to affect refractive stability
* Lid position abnormalities that may affect vision
* Moderate or severe stage glaucoma or optic nerve disease, that would interfere with assessment of or achievement of optimal BCVA
* Visually significant macular disease

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Mean postoperative astigmatism | postoperative 3 months
  Mean postoperative astigmatism

SECONDARY OUTCOMES:
Mean monocular uncorrected distance visual acuity | 3 months postoperatively
  Postoperative mean monocular uncorrected distance visual acuity
Mean monocular corrected distance visual acuity | 3 months postoperatively
  Postoperative mean monocular corrected distance visual acuity

OTHER OUTCOMES:
Percentage of eyes with residual refractive astigmatism within 0.5 D | postoperative 3 months
  Frequency distribution of postoperative refractive astigmatism
Proportion of eyes with uncorrected distance visual acuity 20/x or better | Postoperative 3 months
  Frequency distribution of the proportion of eyes achieving postoperative uncorrected distance visual acuity 20/x or better
Spherical equivalent refractive accuracy | 3 months postoperatively
  Proportion of eyes with postoperative MRSE within 0.50 and 1.00 D

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Rosenthal, MD, Principal Investigator — Kenneth J Rosenthal, MD PC
Locations (1):
- Kenneth J Rosenthal, MD PC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No